CLINICAL TRIAL: NCT01496911
Title: Study to Investigate the Effects of Levocetirizine and Hydroxyzine on Cognitive and Psychomotor Functioning During Simulated Diving at 2 Bar and 4 Bar in Professional Navy Divers
Brief Title: Effects of Levocetirizine and Hydroxyzine on Cognitive and Psychomotor Functioning During Simulated Diving
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Utrecht Institute for Pharmaceutical Sciences (Other)
Collaborators: Royal Netherlands Navy (Unknown)
Responsible Party: Principal Investigator, Dr Joris C Verster, Assistant professor, Utrecht Institute for Pharmaceutical Sciences
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 10-206G/E
Record Dates: First submitted 2011-12-19; First posted 2011-12-21 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Healthy Volunteers
Keywords: Diving; Drugs; Antihistamines; Performance
MeSH Terms: interventions — levocetirizine; Hydroxyzine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Levocetirizine (5 mg) (Experimental)
  Interventions: Drug: Levocetirizine
- Hydroxyzine (50 mg) (Active Comparator)
  Interventions: Drug: Hydroxyzine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levocetirizine — a single oral dose of 5 mg
  Arms: Levocetirizine (5 mg)
Drug: Hydroxyzine — a single oral dose of 50 mg
  Arms: Hydroxyzine (50 mg)
Drug: Placebo — a single oral dose
  Arms: Placebo

SUMMARY:
Antihistamines are commonly used and currently levocetirizine is most frequently prescribed in the Netherlands. They are commonly used by divers, to solve ear, nose and throat problems, especially to open tubal passage. However, the effects of these drugs on cognitive performance have not been investigated during diving.The objective of this study is to investigate the effects of levocetirizine, hydroxyzine and placebo on cognitive and psychomotor functioning during controlled simulated diving in a hyperbaric chamber in professional navy divers at 10 mt (2 bar) and 30 mt (4 bar).It is hypothesized that hydroxyzine will produce significant impairment, and that the magnitude of impairment is related to hyperbaric pressure.

DETAILED DESCRIPTION:
This double-blind, randomized, placebo-controlled cross-over study will comprise of 1 training day and 3 test days. Twenty-four healthy male divers from the Royal Netherlands Navy will participate in this study.The objective of this study is to investigate the single dose effects of levocetirizine (5 mg), hydroxyzine (50 mg) and placebo.

Visit 1 is a training day, and Visit 2-4 are test days. At the test day, subjects receive one of the three medications. One hour after administration of the drugs, subjects will start with the dive in the recompression chamber. After one hour, medication has reached their peak plasma concentration, and effects can be expected. There will be a wash-out period of at least 7 days between the test days.

Subjects will perform one simulated dive at each test day. They first descend in 2 min to a pressure of 4 bar (30 mt), stay for 20 min, the dive continues when they ascend to a pressure of 2 bar (10 mt) with another stay for 20 min. At both depths the 20 min periods are the measuring period to perform the test. At the end they will go to the surface according the decompression profile and stop for 3 min at 9 mt, 8 min at 6 mt and 23 min at 3 mt. These decompression stops are regular for the profile and necessary to prevent decompression sickness.Before and after diving, and at 2 and 4 bar, tests measuring attention, memory, psychomotor, concentration and comprehension ability of the participants are conducted.

ELIGIBILITY:
Inclusion Criteria:

* male healthy volunteer
* He is aged between 18 and 55 years old
* BMI between 18 and 30
* Written informed consent
* Normal static binocular acuity, corrected or uncorrected
* Normal hearing
* Possession of a valid divers certificate and medical fit for diving
* Be considered as reliable and mentally capable of adhering to the protocol.

Exclusion Criteria:

* Female
* Current drug use
* Use of psychoactive medication, including antihistamines
* Prior enrolment in the same study
* Physical or mental illness
* Excessive alcohol use (>21 alcoholic drinks per week)
* Intake of caffeine-containing beverages over 5 glasses per day
* Smoker

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of errors on the cognitive tests | acute (up to 3.5 hours after treatment administration)

SECONDARY OUTCOMES:
Reaction speed on the cognitive tests | acute (up to 3.5 hours after treatment administration)

CONTACTS AND LOCATIONS:
Overall Officials: Joris Verster, PhD, Principal Investigator — Utrecht University
Locations (1):
- Royal Netherlands Navy, Den Helder, North Holland, Netherlands